CLINICAL TRIAL: NCT02306642
Title: Long Term Follow-up of Acute Kidney Injury in Very Low Birth Weight Infants
Brief Title: Follow-up of AKI in Neonates During Childhood Years
Acronym: FANCY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Matthew Harer, MD (Other)
Responsible Party: Sponsor-Investigator, Matthew Harer, MD, Neonatal-Perinatal Medicine Fellow, MD, University of Virginia
Organization: University of Virginia (Other)
Other Study IDs: 17540
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Neonatal Acute Kidney Injury; Childhood Chronic Kidney Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Premature Acute Kidney Injury in NICU: This group of babies born less than 1500 grams will have experienced acute kidney injury based on the modified KDIGO guidelines for acute kidney injury.
- Premature No Acute Kidney Injury in NICU: This group of babies born less than 1500 grams will have not experienced acute kidney injury in the NICU.
- Term No Acute Kidney Injury: This group of babies born at term will have not experienced any acute kidney injury.

SUMMARY:
The purpose of this study is to learn more about how to identify signs of early chronic kidney diseases in children who were born prematurely with low birth weight (less than 3 ½ pounds). Researchers plan to compare the kidney function in children who experienced acute kidney injury (AKI) in the Neonatal Intensive Care Unit (NICU) with those who did not experience it. Evidence from several studies and our experience at UVA show that older children who experienced AKI while in the Pediatric Intensive Care Unit (PICU) have increased risk of developing early chronic kidney disease, and they also show early changes in the urine and blood that is consistent with early chronic kidney disease. In this study, the investigators hope to determine if any of these changes can be detected in early childhood, and if so, at what age we can start detecting these changes.

ELIGIBILITY:
Inclusion Criteria:

* Premature birth for Premature groups
* UVA NICU admission prior to 2 days of life
* Birth weight less than 1500 grams for premature groups
* Premature AKI Study group: Acute Kidney Injury as defined by KDIGO modified criteria during NICU stay at UVA
* Premature no AKI Control group: No AKI during NICU stay
* Term no AKI Control group: No AKI and born at term
* Parental or legal guardian consent obtained

Exclusion Criteria:

- Patients with Congenital Anomalies of the Kidney and Urinary Tract

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born prematurely less than 1500 grams who stayed in the University of Virginia NICU.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Composite Abnormality | Age 2-7 years
  Either eGFR > 90, urine protein/creatinine > 0.2, or BP > 95th percentile for age and height

SECONDARY OUTCOMES:
Growth | Age 2-6 years
  Evaluation of height, weight and BMI
Kidney Size | Age 2-6 years
  Evaluation of kidney size
Urinary Biomarkers | Age 2-6 years
  Evaluation of urine for biomarkers which can be used to detect early chronic kidney disease

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States